CLINICAL TRIAL: NCT00982254
Title: A Comparison of the Pharmacodynamic and Pharmacokinetic Properties of Oral Insulin vs. s.c. Regular Insulin in Type 2 Diabetic Patients
Brief Title: Oral Insulin: A Comparison With Subcutaneous Regular Human Insulin in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Profil Institut für Stoffwechselforschung GmbH (Industry)
Collaborators: Emisphere Technologies, Inc. (Industry)
Responsible Party: Tim Heise, MD, Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 175A-C-02
Record Dates: First submitted 2009-09-14; First posted 2009-09-23 (Estimated); Last update posted 2009-09-23 (Estimated); Status verified 2009-09

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; Oral Insulin; Pharmacokinetics; Pharmacodynamics
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral Insulin (Experimental): oral insulin capsule formulation
  Interventions: Drug: Oral insulin
- Subcutaneous Insulin (Active Comparator): Subcutaneous injection of regular human insulin
  Interventions: Drug: regular human insulin

INTERVENTIONS:
Drug: Oral insulin — oral insulin capsule formulation (150 U insulin/200 mg 4-CNAB in one capsule); single dose administration of 300 U insulin (in two capsules) and of 150 U insulin (one capsule) on two separate dosing days.
  Arms: Oral Insulin
Drug: regular human insulin — subcutaneous injection of 15 U regular human insulin; single dose administration on one separate dosing visit.
  Other Names: Humulin R (100 U/mL)
  Arms: Subcutaneous Insulin

SUMMARY:
This study compared the pharmacokinetic and pharmacodynamic properties of an oral insulin formulation with that of a standard subcutaneous injection of regular human insulin.

DETAILED DESCRIPTION:
This study was a single centre, randomized, 3-period crossover study performed in patients with type 2 diabetes. Patients received single doses of an oral insulin formulation and subcutaneous regular human insulin on separate visits.

The primary objective of this study was to compare the pharmacokinetic and pharmacodynamic properties of an oral insulin formulation with that of 15 U subcutaneous injected regular human insulin.

Pharmacokinetic and pharmacodynamic parameters including bioavailability and bioefficacy were measured during 6-hour glucose clamp experiments.

Study duration: 2 months

ELIGIBILITY:
Inclusion Criteria:

* Male subjects between the ages of 35 and 70 years, inclusive, with Type 2 diabetes mellitus as defined by the ADA criteria for more than one year
* Subjects must have Body Mass Index (BMI) < 36 kg/m²
* Stable glycemic control (HbA1C <11%)
* Subjects must be off all oral hypoglycemic agents 24 hours prior to each study dosing day and off any investigational drug for at least 4 weeks
* Subjects must refrain from strenuous physical activity beginning 72 hours prior to admission and through the duration of the study
* Subjects must be willing and able to be confined to the Clinical Research Unit as required by the protocol
* Subjects must be willing and able to provide written informed consent

Exclusion Criteria:

* History or presence of clinically significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, neurological or infectious disorders capable of altering the absorption, metabolism or elimination of drugs, or of constituting a risk factor when taking the study medication
* Subjects with gastroparesis, orthostatic hypotension and hypoglycemia unawareness (autonomic neuropathy).
* Subjects with "brittle" diabetes or predisposition to severe hypoglycemia, e.g., 2 or more serious hypoglycemic episodes (requiring another's assistance) within the past year, or any hospitalization or emergency room visit due to poor diabetic control within the past 6 months.
* Evidence of significant active hematological disease and/or cumulative blood donation of 1 unit (500 mL) or more including blood drawn during clinical trials in the last 3 months
* Positive hepatitis B (hepatitis B surface antigen) and/or hepatitis C (hepatitis C antibody) serology
* Positive HIV serology
* Evidence of significant active neuropsychiatric disease
* Known allergy to human insulin excipients contained in these products
* Regular alcohol intake greater than 28 units*/week (male), or 21 units/week (female), or subjects unwilling to stop alcohol for the duration of the study (* 1 unit = 8 g ethanol, ¼ liter of beer or 1 glass wine or 1 measure of spirits)
* Intake of any drug which in the evaluation of the investigator may interfere with the interpretation of trial results or are known to cause clinically relevant interference with insulin action, glucose utilisation or recovery from hypoglycaemia.
* Treatment with s.c. insulin injections.
* Investigators, site personnel directly affiliated with this study, and their immediate families. Immediate family is defined as a spouse, parent, child or sibling, whether biological or legally adopted
* Have any other condition (including drug abuse, alcohol abuse, or psychiatric disorder) that, in the opinion of the investigator, precludes the patient from following and completing the protocol.

Ages: 35 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2001-10; Primary Completion 2001-11 (Actual)

PRIMARY OUTCOMES:
Glucose Infusion Rate (GIR) | For each treatment continuously from 6 hours before dosing until 6 hours after dosing

SECONDARY OUTCOMES:
Plasma insulin concentration | For each treatment at regular times from 6 hours before dosing until 6 hours after dosing
Plasma C-Peptide | For each treatment at regular times from 6 hours before dosing until 6 hours after dosing
Adverse Events | For each treatment before and after end of clamp

CONTACTS AND LOCATIONS:
Overall Officials: Tim Heise, MD, Principal Investigator — Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany

REFERENCES:
- [Derived] Kapitza C, Zijlstra E, Heinemann L, Castelli MC, Riley G, Heise T. Oral insulin: a comparison with subcutaneous regular human insulin in patients with type 2 diabetes. Diabetes Care. 2010 Jun;33(6):1288-90. doi: 10.2337/dc09-1807. Epub 2010 Feb 25. PMID 20185734